CLINICAL TRIAL: NCT01967407
Title: Prospective, Monocentric, Clinical Phase-I/II Study of the Effectiveness of the Percutaneous Irreversible Electroporation (IRE) of Locally Confined Kidney Tumors (Renal Cell Carcinomas).
Brief Title: IReversible Electroporation of Kidney Tumors Before Partial Nephrectomy.
Acronym: IRENE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Magdeburg (Other)
Responsible Party: Principal Investigator, Johann J. Wendler, MD, Dr. med., University of Magdeburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DE-UKMD-URO-001; DRKS00004266 (Other: DRKS (German Clinical Trials Registry)); U1111-1140-0415 (Other: Universal Trial Number (UTN)); DRKS00004266 (Other: Internat. Clinical Trials Registry Platform ICTRP, WHO); EUDAMED-No.: CIV-12-04-006021 (Other: BfArM, German Federal Inst. for Drugs & Medical Devices); 00020520 (Other: DIMDI, German Inst. for Med. Documentation & Information)
Record Dates: First submitted 2013-10-15; First posted 2013-10-22 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Kidney Tumor; Renal Cell Cancer
Keywords: kidney tumor; renal cell cancer; RCC; irreversible electroporation; IRE; partial kidney resection; percutaneous; ablation; IRENE
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Electroporation; Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- renal tumor <4cm, suspected RCC (Experimental): Intervention/ Time point: Irreversible Electroporation at day 0 of each patient.
  Interventions: Procedure: Irreversible Electroporation (IRE)

INTERVENTIONS:
Procedure: Irreversible Electroporation (IRE) — Percutaneous CT-fluoroscopic-guided Irreversible Electroporation.
  Other Names: NanoKnife (Tissue Ablation) System, AngioDynamics Inc.

SUMMARY:
The aim of the study is the evaluation of the ablation efficiency of the percutaneous irreversible electroporation (IRE) as primary ablation therapy of locally confined renal cell carcinoma (≤4cm, see inclusion and exclusion criteria).

The ablation success will be proofed by magnet resonance imaging (MRI) and histologically after partial kidney resection or nephrectomy 4 weeks after IRE. Hypotheses: Kidney tumors ≤4cm can be ablated completely by percutaneous IRE. Surrounded structures and renal tissue can be preserved.

DETAILED DESCRIPTION:
Health Condition or Problem studied:

1. International Statistical Classification of Diseases and Related Health Problems, Tenth Revision (ICD10): C64 - Malignant neoplasm of kidney, except renal pelvis
2. ICD10: D41.0 - Neoplasm of uncertain or unknown behaviour: Kidney

Interventions/Observational Groups Arm 1:

1. Initial diagnostical examination of the renal mass.
2. If any extended diagnostical examination for treatment planning.
3. Day -29 to -1: Recruitment.
4. Day -1: MRI of the kidney, Karnofsky, physical examination, blood chemistry, urosonography, if any renal scintigraphy, life quality assessment.
5. Day 0: Percutaneous diagnostical biopsy with histopathological investigation and therapeutically, CT- and/or ultrasound-guided, ECG-synchronized irreversible electroporation (IRE) of the kidney tumor in endotracheal anaesthesia und muscle relaxation. Use of 1-6 IRE probes with 90-100 pulses of 1500-3000 volts und 20-50 amperes each.
6. Day 1-7: Postinterventional follow-up: MRI of the kidneys, Karnofsky, physical examination, blood chemistry, urosonography, life quality assessment.
7. Day 27: Postinterventional follow-up: MRI of the kidneys, Karnofsky, physical examination, blood chemistry, urosonography, if any renal scintigraphy, life quality assessment.
8. Day 28: Open surgery partial kidney resection or tumor nephrectomy of the IRE treated kidney resp. kidney tumor region with histopathological investigation.
9. Day 29-37: Postoperative follow-up: physical examination, blood chemistry, urosonography, life quality assessment.
10. Day 112: Study-Follow-up: MRI of the kidneys, Karnofsky, physical examination, blood chemistry, urosonography, if any renal scintigraphy, life quality assessment. Termination of the study.
11. Study closed, Individual follow-up due to the European Association of Urology guideline.

Recruitment:

* (Anticipated or Actual) Date of First Enrollment: 2013/10/14
* Planned/Actual: Opened
* Target Sample Size: 20
* Monocentric/Multicentric trial: Monocentric trial
* National/International: National

ELIGIBILITY:
Inclusion Criteria:

* one or more localized, resectable kidney tumors (≤4 cm) suspicious of malignancy or histology -proven renal cell cancer (RCC)
* patients desire for therapy and surgical therapy
* Karnofsky-index >70%
* Age ≥ 18 years
* life expectancy ≥ 12 month
* compliance of the patient taking part in a study
* informed consent

Exclusion Criteria:

* violation against one or more inclusion criteria
* cardial pacemaker or other electrical implants
* QT-interval >550 ms or cardiac arrhythmias or condition after myocardial infarction, that make an ECG-synchronisation unfeasible
* known cardial ejection fraction < 30% or NYHA III or III-IV
* known epilepsy
* second malignancy (except basal-cell carcinoma and cervical carcinoma in situ)
* immunosuppression or HIV-positive patients
* active infection or severe health interference, that make taking part in a study unfeasible
* pregnancy, lactation period, no contraception
* metastatic disease
* palliative status
* running or executed RCC therapy
* taking part in another clinical study for RCC
* inoperable
* rejection of interventional or surgical therapy by the patient
* circulatory instability
* general contraindications for anesthesia, endotracheal anesthesia and muscle relaxation
* psychiatric disorders that make taking part in a study or giving informed consent unfeasible
* haemorrhage, impossible intermission of taking blood thinner, untreatable thrombophilia
* thromboplastin time ≤50 %, thrombocytes ≤50 Gpt/L; partial thromboplastin time >50
* MRI incompatibility
* metal implants <1 cm closed to the kidney / kidney tumor
* contraindication for biopsy and punction of the renal tumor under CT-guidance
* untreated urinary retention
* renal pelvis tumor, suspected transitional cell cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
analysis of ablation effectiveness of non-metastatic renal tumors <4cm 28 days by after irreversible electroporation (NanoKnife, AngioDynamics Inc.) by histopathological examination of partial kidney resection specimens | 28 days
  onco-therapeutic effectiveness, measured against persistent active tumor / cancer cells by histopathological and magnet resonance imaging analysis

SECONDARY OUTCOMES:
safety | 4 month
  * adverse effects
  * Assessment of the procedural compliance
  * Assessment of the Quality of Life (QoL)

CONTACTS AND LOCATIONS:
Overall Officials: Uwe- B. Liehr, Dr. med., Principal Investigator — Department of Urology, University Magdeburg, Germany.; Martin Schostak, Prof. Dr., Study Director — Department of Urology, University Magdeburg, Germany; Johann J. Wendler, Dr. med., Principal Investigator — Department of Urology, University Magdeburg, Germany
Locations (4):
- Germany (4):
  - Department of Pathology University Hospital Otto-von-Guericke-University Magdeburg, Magdeburg, Saxony-Anhalt
  - Department of Radiology University Hospital Otto-von-Guericke-University Magdeburg, Magdeburg, Saxony-Anhalt
  - Department of Urology University Hospital Otto-von-Guericke-University Magdeburg, Magdeburg, Saxony-Anhalt
  - MVZ Hanse Histologikum GmbH Hamburg, Hamburg

REFERENCES:
- [Background] Liehr UB, Wendler JJ, Blaschke S, Porsch M, Janitzky A, Baumunk D, Pech M, Fischbach F, Schindele D, Grube C, Ricke J, Schostak M. [Irreversible electroporation: the new generation of local ablation techniques for renal cell carcinoma]. Urologe A. 2012 Dec;51(12):1728-34. doi: 10.1007/s00120-012-3038-8. German. PMID 23139026
- [Background] Jiang C, Davalos RV, Bischof JC. A review of basic to clinical studies of irreversible electroporation therapy. IEEE Trans Biomed Eng. 2015 Jan;62(1):4-20. doi: 10.1109/TBME.2014.2367543. PMID 25389236
- [Derived] Wendler JJ, Porsch M, Fischbach F, Pech M, Schostak M, Liehr UB. Letter to the Editor Concerning "Irreversible Electroporation (IRE) Fails to Demonstrate Efficacy in a Prospective Multicenter Phase II Trial on Lung Malignancies: The ALICE Trial" by Ricke et al. 2015 (doi:10.1007/s00270-014-1049-0). Cardiovasc Intervent Radiol. 2015 Aug;38(4):1064-5. doi: 10.1007/s00270-015-1096-1. Epub 2015 Apr 23. No abstract available. PMID 25902855
- See also: Department of Urology, University Magdeburg — http://urologie.med.uni-magdeburg.de/urologie.html